CLINICAL TRIAL: NCT01676337
Title: A Text-message Appointment Reminder System to Improve Patient Adherence With Outpatient Follow-up Appointments
Brief Title: Text Message Appointment Reminders
Acronym: TAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sanjay Arora, MD, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-12-00239
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Text Messages; Emergencies
Keywords: Text messaging; Clinic appointment attendance; Emergency department; Primary care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients randomized to the control arm will not receive text message reminder regarding their upcoming appointment.
- Text message appointment reminder (Experimental): Patients randomized to the intervention arm will receive text message appointment reminders including date, time, and location seven, three and one day prior to their scheduled clinic appointments. All appointment reminders will then be delivered automatically.
  Interventions: Other: Text message appointment reminder

INTERVENTIONS:
Other: Text message appointment reminder — Patients randomized to the intervention arm will receive text message appointment reminders including date, time, and location seven, three and one day prior to their scheduled clinic appointments. All appointment reminders will then be delivered automatically.
  Arms: Text message appointment reminder

SUMMARY:
This project proposes administer and evaluate via a randomized controlled trail a text message-based appointment reminder system to promote attendance at clinic appointments after ED discharge.

DETAILED DESCRIPTION:
Failure to attend scheduled clinic appointments causes inefficiency within the healthcare system, and frequently results in ED visits for non-emergent conditions such as medication refills, ambulatory care sensitive conditions which are potentially preventable with appropriate outpatient management (e.g. foot infections). Many patients seen in the ED report they were unaware of past or future outpatient appointments for which they had been scheduled. These patients are clearly in need of primary care, yet fail to attend 30% of all scheduled outpatient appointments. Patients most often report that they failed to attend scheduled appointments as a result of forgetfulness or confusion regarding dates, times, or locations. National data confirmed by our previous work in the LAC+USC ED demonstrates that > 80% of this population reports using a text-capable mobile device. The investigators believe a system of text message appointment reminders has tremendous potential to facilitate clinic attendance among these patients in desperate need of primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Able to provide consent and read in English or Spanish
* Have a text message capable mobile phone
* Know how to receive text messages
* Have upcoming scheduled clinic appointments

Exclusion Criteria:

* Unable to provide written informed consent
* Incarcerated
* Critically ill
* Altered Mental Status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Adherence with scheduled appointments within 30 days post-enrollment | 30 days

SECONDARY OUTCOMES:
Adherence with scheduled appointments within 6 months post-enrollment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Arora, MD, Principal Investigator — University of Southern California; Michael Menchine, MD, MPH, Principal Investigator — University of California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Arora S, Burner E, Terp S, Nok Lam C, Nercisian A, Bhatt V, Menchine M. Improving attendance at post-emergency department follow-up via automated text message appointment reminders: a randomized controlled trial. Acad Emerg Med. 2015 Jan;22(1):31-7. doi: 10.1111/acem.12503. Epub 2014 Nov 11. PMID 25388481